CLINICAL TRIAL: NCT03855085
Title: Assessment of the Reproducibility of Kidney Transplant Sonographic Volume Measurement
Brief Title: Kidney Transplant Volumetry
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19-Volumetrie GreffeR
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Kidney Transplant; Complications
Keywords: Kidney transplant; volumetry; ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study assesses the reproducibility of 3 different formulas in calculating the volume of a transplanted kidney by ultrasound in-vivo measurements.

3 series of measurements will be performed by 2 different operators during the usual ultrasound follow-up of the renal transplant.

DETAILED DESCRIPTION:
The 3 series of measurements

1. Longitudinal section: maximum longitudinal length, width at the hilum, maximum width, width at the upper third, longitudinal cross-sectional area
2. Transverse section at the hilum : thickness, width, hilar cross-sectional area
3. Largest transverse section : thickness, width, maximum transverse cross-sectional area

Clinical and biological patient data collection:

age, gender, date of transplantation, serum creatinine and glomerular filtration rate (GFR), kidney transplant placement (right or left iliac fossa), acute illness or usual follow-up

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recepients with ultrasound follow-up at the University Hospital of Tours
* Age more than 18 years old

Exclusion Criteria:

* Renal deformity of extrinsic origin
* Early post-transplant period (first 3 days post-transplant)
* Transplanted organ out of the field of view
* Dual kidney transplant
* Opposition to the data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Intraclass coefficient of correlation of the ultrasound volume measurement | 6 months
  The inter-observer and intra-observer variability of the ultrasound volume measurement of the kidney graft will be assessed using the intraclass coefficient of correlation (ICC)

SECONDARY OUTCOMES:
Intraclass coefficient of correlation of the volume formula parameters. | 6 months
  The reproducibility of each formula parameter will also be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Gradinaru, Tours, France

IPD SHARING:
Plan to Share IPD: No